CLINICAL TRIAL: NCT04175106
Title: Establishing Optimal Nutritional Quality of Blueberries: a Proof of Concept Study to Improve the Nutritional Quality of the Average Diet Using Common Plant Breeding and Processing Practices.
Brief Title: Evaluating the Availability of Berry Phytonutrients Post-consumption of Fresh and Processed Blueberry by Healthy Adults
Acronym: BAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Carolina State University (Other)
Collaborators: Foundation for Food and Agriculture Research (Unknown)
Responsible Party: Principal Investigator, Colin D. Kay, Associate Professor in Nutrition Science, PhD, North Carolina State University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 19138
Record Dates: First submitted 2019-11-13; First posted 2019-11-22 (Actual); Results first posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- a phytochemical-rich blueberry variety (Experimental): Single-time consumption of 150 g phytochemical-rich blueberry per participant.
  Interventions: Other: a non-traditional (i.e., not typically available in the supermarket) blueberry cultivar bred using natural plant breeding techniques and established as having enhanced nutritive value
- a phytochemical-poor blueberry variety (Experimental): Single-time consumption of 150 g phytochemical-poor blueberry per participant.
  Interventions: Other: a standard commercially available blueberry variety (i.e., cultivar)
- a "minimally processed" blueberry-rich protein bar (Experimental): Single-time consumption of blueberry-rich protein bar matched for 150 g blueberry phytochemicals.
  Interventions: Other: a "minimally processed" blueberry-rich protein bar
- a blueberry control beverage of matched-nutritive content (Placebo Comparator): Single-time consumption of control beverage matched for the macronutrient content of the blueberry-rich protein bar.
  Interventions: Other: a control beverage of matched-nutritive content

INTERVENTIONS:
Other: a non-traditional (i.e., not typically available in the supermarket) blueberry cultivar bred using natural plant breeding techniques and established as having enhanced nutritive value — 150 g of a non-traditional (i.e., not typically available in the supermarket) blueberry cultivar bred using natural plant breeding techniques and established as having enhanced nutritive value.
  Dietary restrictions will be observed (i.e. avoidance of food or supplements containing berry phytonutrients) for 7 days before each arm visit and throughout the study days.
  Arms: a phytochemical-rich blueberry variety
Other: a standard commercially available blueberry variety (i.e., cultivar) — 150 g of a standard commercially available blueberry variety (i.e., cultivar).
  Dietary restrictions will be observed (i.e. avoidance of food or supplements containing berry phytonutrients) for 7 days before each arm visit and throughout the study days.
  Arms: a phytochemical-poor blueberry variety
Other: a "minimally processed" blueberry-rich protein bar — A "minimally processed" blueberry-rich protein bar matched to the phytonutrient content of the 150 g of the non-traditional blueberry.
  Dietary restrictions will be observed (i.e. avoidance of food or supplements containing berry phytonutrients) for 7 days before each arm visit and throughout the study days.
  Arms: a "minimally processed" blueberry-rich protein bar
Other: a control beverage of matched-nutritive content — The matched nutritive content of the blueberry-rich protein bar will be dissolved in whey protein
  Dietary restrictions will be observed (i.e. avoidance of food or supplements containing berry phytonutrients) for 7 days before each arm visit and throughout the study days.
  Arms: a blueberry control beverage of matched-nutritive content

SUMMARY:
This study will evaluate the availability of phytonutrients in two blueberry varieties, chosen for their phytonutrient levels. This will be compared to phytonutrient-matched processed protein bar and a macronutrient-matched control meal, in healthy human volunteers. Blueberry phytonutrients will be analyzed in blood and urine over a four-day period, 48h prior to consumption and 48h after. The participants will consume each of the four meals over a 3-month period (4-way crossover design, 4 blocks of 4-day periods). The main objective of this study is to compare the proportions of blueberry phytonutrients recovered in the blood and urine after ingestion of the four treatments. We hypothesize that phytonutrient content will be predictive of human bioavailability and that a berry-enriched processed product will have similar phytonutrient bioavailability to unprocessed berries.

The results of this study may establish if the nutritional value of a berry can be predicted or enhanced to provide elevated nutritional quality, with the ultimate goal of maximizing the health benefits of fruit consumption. As it is challenging for many to increase their fruit and vegetable intake to government recommended levels (5+ servings per day), the present proof-of-concept study explores a reasonable approach to help consumers achieve optimal health associated with high fruit and vegetable intakes, within the context of current consumption patterns, through enhancement of the nutritional density and bioavailability of common fruits and consumer products.

DETAILED DESCRIPTION:
This study will evaluate the availability of phytonutrients in two blueberry varieties, chosen for their phytonutrient levels. This will be compared to phytonutrient-matched processed protein bar and a macronutrient-matched control meal, in healthy human volunteers. Blueberry phytonutrients will be analyzed in blood and urine over a four-day period, 48h prior to consumption and 48h after. The participants will consume each of the four meals over a 3-month period (4-way crossover design, 4 blocks of 4-day periods).

The main objective of this study is to compare the proportions of blueberry phytonutrients recovered in the blood and urine after ingestion of the four treatments.

After eligibility is confirmed, subjects will be randomly assigned to the four berry related interventions. The consumption of each intervention corresponds to one study period, which are separated by one-week washout. Blood will be collected at baseline and across 48h (1h, 3h, 6h, 9h, 24h, 48h) after intervention consumption while urine will be collected for 48h before and after intervention (-48h, -24h, 0-9h, 9-24h, 24-48h).

ELIGIBILITY:
Inclusion Criteria:

* male and female adults between 25-65 years;
* non-smokers, non-tobacco users (no vaping nor deeping), or who ceased it ≥ 6 months ago;
* who present no allergies to fruits or vegetables containing polyphenolic (e.g. anthocyanins, flavonoids) and phenolic acids such as blueberries, red apple, strawberry, red orange, purple onion and broccoli;
* who present no allergies to dairy products, specifically whey protein, fructose or salicylates;
* who are generally healthy and without chronic diseases including cancer, type 1 and 2 diabetes;
* who are not prescribed thyroid or hypoglycemic medication or hormone replacement therapy (HRT) (due to the likely concomitant effects that these medications cause on the primary endpoint in the trial);
* who has not been consuming any phytonutrient-containing supplements (e.g. with cocoa, coffee, berry, polyphenol, flavonoid, or anthocyanin extracts) for at least a month before the study and willing to not consume it during the study;
* who lives within 40 miles from the North Carolina Research Campus (NCRC) campus;
* those agreeing to restrict dietary intake of rich sources of phytonutrients targeted on the study during the wash-out and clinical sampling periods, agreeing to comply with a biological sampling protocol involving the collection of urine and blood samples, and to record their additional dietary intake over 2 days before each intervention, and two days after the intake of the intervention treatments;
* who have BMI ≥18.5 and ≤ 30 (lbs/in2x703);
* who have a successful (i.e., within normal range for healthy individuals) biochemical, hematological and urine analyses assessed by the clinical advisor as established during the screening period prior to final enrollment.

Exclusion Criteria:

* current smokers (vaping and deeping included), or ex-smokers ceasing < 6 months before recruitment;
* pregnant or breastfeeding;
* subjects with existing or significant past medical history of vascular disease or medical conditions likely to affect the study measures i.e. vascular disease, circulatory (i.e. Reynaud's), diabetes, hepatic, renal, digestive, hematological, cancer, or thyroid disease;
* fructose intolerant subjects or those with known allergy to salicylates, dairy products, specifically whey protein, or to berries;
* those unprepared to adhere to dietary restrictions for 1 week preceding and during each intervention or unwilling to comply with the assessments per protocol;
* who are in parallel participation in another research project involving dietary intervention and/or sampling of biological fluids/material;
* those on therapeutic diets or having experienced substantial weight loss (to be judged by clinical advisor) within 3 months of screening;
* those taking phytonutrient-containing supplements (e.g. with cocoa, coffee, berry, polyphenol, flavonoid, or anthocyanin extracts), unwilling to cease intake during, and 1 month preceding the trial, or unwilling to stop existing intake of other supplements or regular use of large-dose nutrient, herbal, and dietary supplements during the past one to two weeks, or planning to use them during the study;
* prescribed thyroid, hypoglycemic medication or HRT medication -other medications will be assessed for suitability by the clinical advisor;
* those having donated blood in the last month;
* individuals that consume more than 1 and 2 drinks of alcohol per day for women and men, respectively, or more than 7 and 14 drinks per week for women and men, respectively (U.S. Department of Health and Human Services and U.S. Department of Agriculture Dietary guidelines 2015-2020);
* currently on a weight-reducing plan or using weight-loss medications (e.g., selective serotonin reuptake inhibitors, steroids, Ritalin, appetite suppressants such as Diethylpropion or Amfepramone, and weight loss medications such as Alli, Xenical, Qsymia, Belviq, Contrave, and Saxenda), or planning to continue this treatment during the 10-week period of the study;
* who has BMI<18.5 and >30 (lbs/in2x703);
* who presents abnormal biochemical, hematological or urinary results, and measurements considered to be counter-indicative for the study, including: kidney and liver function, fasting glucose (especially if indicative of diabetes), lipid abnormalities, full blood count as established during the screening period prior to final enrollment.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colin D Kay, PhD, Principal Investigator — North Carolina State University
Locations (1):
- Plants for Human Health Institute, North Carolina State University, Kannapolis, North Carolina, United States

REFERENCES:
- [Result] Santana MC, Rathore AS, Chandra P, Everhart JL, Schulz H, Granillo CD, Ferruzzi MG, Iorizzo M, Lila MA, Diaz JT, Kay CD. Bioavailability and pharmacokinetics of (poly)phenols following consumption of selected blueberries and a blueberry-rich protein bar by adult males and females: a randomized, crossover, controlled trial. Am J Clin Nutr. 2025 Apr;121(4):779-794. doi: 10.1016/j.ajcnut.2025.01.028. Epub 2025 Jan 31. PMID 39894303
- See also: Publication of Clinical Study Results — https://doi.org/10.1016/j.ajcnut.2025.01.028

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 75 participants were recruited and screened from the local community surrounding the North Carolina Research Campus, Kannapolis, North Carolina, between December 2019 and July 2021. Clinical screening and interventions were conducted at the Human Research Core at the Nutrition Research Institute (University of North Carolina-Chapel Hill). The trial was completed in October 2021.
Pre-assignment Details: 29 out of 75 screened participants were enrolled into the study and randomized to interventions. Of those not enrolled, 20 participants did not meet inclusion criteria, 17 declined to participate and 9 did not follow up.
Groups:
- Phytochemical-rich and -Poor Blueberry Varieties, Blueberry-rich Protein Bar and a Control Beverage: All enrolled study participants were assigned to 13 distinct randomized intervention sequences where they consumed the following interventions, one at a time, and separated by 30.0±40.6 d of compliance break then 1-week of washout period: 150 g of a Phytochemical-rich Blueberry Variety (Elliott Blueberry Variety), 150 g of a Phytochemical-poor Blueberry Variety (Olympia Blueberry Variety), a "Minimally Processed" Blueberry-rich Protein Bar matched to the phytonutrient content of the 150 g of Phytochemical-rich Blueberry Variety, and a Blueberry Control Beverage of Matched-nutritive Content in a randomized order.
Period: Overall Study
Arm/Group | Phytochemical-rich and -Poor Blueberry Varieties, Blueberry-rich Protein Bar and a Control Beverage
Started | 29
Phytochemical-rich Blueberry Variety | 18
Phytochemical-poor Blueberry Variety | 23
"Minimally Processed" Blueberry-rich Protein Bar | 22
Blueberry Control Beverage of Matched-nutritive Content | 23
Completed | 18
Not Completed | 11
Not completed — Discontinued intervention (COVID-19) | 2
Not completed — Non-compliance | 3
Not completed — Lost to Follow-up | 1
Not completed — Lack of Availability | 3
Not completed — Discomfort | 2

BASELINE CHARACTERISTICS:
Population: Baseline data shown from baseline visits of participants who completed participation in the study across all four arms/groups (i.e., 18 participants).
Arm/Group | Phytochemical-rich and -Poor Blueberry Varieties, Blueberry-rich Protein Bar and a Control Beverage
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.06 (12.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 18
Systolic Blood pressure, mmHg [Mean (Standard Deviation); unit: mmHg] | 116.12 (13.00)
Diastolic Blood pressure, mmHg [Mean (Standard Deviation); unit: mmHg] | 71.54 (7.63)
BMI, kg/m2 [Mean (Standard Deviation); unit: kg/m2] | 24.75 (2.99)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 73.8 (13.72)
Height (m) [Mean (Standard Deviation); unit: meter] | 1.72 (0.10)

OUTCOME MEASURES:

1. Primary Outcome: Total Urinary Recovery of (Poly)Phenolic Metabolites Across Treatments
Description: Concentration of 185 (poly)phenolic metabolites in urine was measured after consumption of the treatments using broad spectrum metabolomic analysis via UPLC-MS/MS (ultra-performance liquid chromatography coupled with tandem mass spectrometry). Recovery of each metabolite was calculated by multiplying the concentration of the metabolite (ng/mL) by the volume of urine (mL) in each collection then converted to milligrams. The total urinary recovery of each (poly)phenolic metabolite was assessed as a measurement of their bioavailability, and it was established as the sum of the recovery from each urine collection (0 h to 48 h postintervention) minus the mean of the 48 h and 24 h baseline collections per participant and treatment. Then, it was averaged across participants per treatment and per metabolite, and further summed across metabolites. Therefore, data reported for each treatment represents the sum of the means of total urinary recovery across (poly)phenolic metabolites.
Time Frame: 4 days of urine collection per intervention; -48, -24, 0-9, 9-24 and 24-48 hours collections of urine.
Population: All participants who completed all study visits. This analysis was pre-specified to only report data for (poly)phenolic metabolites that displayed treatment effects (p < 0.05) in cumulative urinary excretion (i.e., 22 (poly)phenolic metabolites). Sum of the means of total urinary recovery across metabolites is reported per treatment.
Measure: Number; unit: mg
Groups:
- Phytochemical-rich Blueberry Variety (Elliott Blueberry Variety): Single-time consumption of 150 g of a Phytochemical-rich Blueberry Variety (Elliott Blueberry Variety) in a randomized order, and separated by 30.0±40.6 d of compliance break then 1-week of washout period from other interventions.
- Phytochemical-poor Blueberry Variety (Olympia Blueberry Variety): Single-time consumption of 150 g of a Phytochemical-poor Blueberry Variety (Olympia Blueberry Variety) in a randomized order, and separated by 30.0±40.6 d of compliance break then 1-week of washout period from other interventions.
- "Minimally Processed" Blueberry-rich Protein Bar: Single-time consumption of a "Minimally Processed" Blueberry-rich Protein Bar matched to the phytonutrient content of the 150 g of Phytochemical-rich Blueberry Variety in a randomized order and separated by 30.0±40.6 d of compliance break then 1-week of washout period from other interventions.
- Control Beverage of Matched-nutritive Content: Single-time consumption of a control beverage matched for the macronutrient content of the blueberry-rich protein bar in a randomized order and separated by 30.0±40.6 d of compliance break then 1-week of washout period from other interventions.
Arm/Group | Phytochemical-rich Blueberry Variety (Elliott Blueberry Variety) | Phytochemical-poor Blueberry Variety (Olympia Blueberry Variety) | "Minimally Processed" Blueberry-rich Protein Bar | Control Beverage of Matched-nutritive Content
Number analyzed (Participants) | 18 | 18 | 18 | 18
mg | 179.50 | 142.41 | 127.78 | 83.15
Statistical Analysis 1: Comparison: Phytochemical-rich Blueberry Variety (Elliott Blueberry Variety) vs Phytochemical-poor Blueberry Variety (Olympia Blueberry Variety) vs "Minimally Processed" Blueberry-rich Protein Bar vs Control Beverage of Matched-nutritive Content; This study was powered to detect a 25% change in total urinary (poly)phenolic metabolites at 80% power and α = 0.05 based on means and effect sizes published in previous (poly)phenol bioavailability studies that applied crossover or parallel design; Test type: Other; p < 0.05, ANOVA — Concentration data was assessed for normalization using the Shapiro-Wilk test and normalized using log(1+x) when deemed non-normalized; Changes across groups via linear mixed-effects repeated measures ANOVA, and post-hoc analysis (Bonferroni test and Kenward-Roger degrees of freedom)

2. Primary Outcome: Serum Area Under the Curve (AUC) of (Poly)Phenolic Metabolites Across Treatments
Description: Concentration of 185 (poly)phenolic metabolites in blood was measured after consumption of the treatments using broad spectrum metabolomic analysis via UPLC-MS/MS (ultra-performance liquid chromatography coupled with tandem mass spectrometry). The area under the curve (AUC) of each (poly)phenolic metabolite in serum was assessed as a measurement of the bioavailability of these metabolites per participant and treatment. It was calculated using concentration and time data in the software Phoenix WinNonlin (version 8.3, Certara). Then, AUC was averaged across participants per treatment and per metabolite, and the mean AUCs were further summed across metabolites. Therefore, data reported for each treatment represents the sum of the means of AUC across (poly)phenolic metabolites.
Time Frame: 3 days of blood collection per intervention; 1 baseline collection, followed by 1, 3, 6, 9, 24 and 48 hours post-treatment collections of blood.
Population: All participants who completed all study visits. This analysis was pre-specified to only report data for (poly)phenolic metabolites that displayed treatment-by-time, treatment, and time effects (p < 0.05) in serum concentration (i.e., 20 (poly)phenolic metabolites). Sum of the means of AUC across metabolites is reported per treatment.
Measure: Number; unit: ng*h/mL
Arm/Group | Phytochemical-rich Blueberry Variety (Elliott Blueberry Variety) | Phytochemical-poor Blueberry Variety (Olympia Blueberry Variety) | "Minimally Processed" Blueberry-rich Protein Bar | Control Beverage of Matched-nutritive Content
Number analyzed (Participants) | 18 | 18 | 18 | 18
ng*h/mL | 3889.34 | 3049.40 | 3515.23 | 2704.96
Statistical Analysis 1: Comparison: Phytochemical-rich Blueberry Variety (Elliott Blueberry Variety) vs Phytochemical-poor Blueberry Variety (Olympia Blueberry Variety) vs "Minimally Processed" Blueberry-rich Protein Bar vs Control Beverage of Matched-nutritive Content; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.05, ANOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Maximum Serum Concentration [Cmax] of (Poly)Phenolic Metabolites Between the Treatments
Description: Concentration of 185 (poly)phenolic metabolites in serum was measured after consumption of the treatments using broad spectrum metabolomic analysis via UPLC-MS/MS (ultra-performance liquid chromatography coupled with tandem mass spectrometry). The maximum serum concentration [Cmax] of each (poly)phenolic metabolite in serum was calculated per participant and treatment using concentration and time data in the software Phoenix WinNonlin (version 8.3, Certara). Then, it was averaged across participants per treatment and per metabolite, and further averaged across metabolites. Therefore, data reported for each treatment represents the mean of the means of Cmax across (poly)phenolic metabolites.
Time Frame: as for outcome 2
Population: All participants who completed all study visits. This analysis was pre-specified to only report data for (poly)phenolic metabolites that displayed treatment-by-time, treatment, and time effects (p < 0.05) in serum concentration (i.e., 20 (poly)phenolic metabolites). Mean of the means of Cmax across metabolites is reported per treatment.
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | Phytochemical-rich Blueberry Variety (Elliott Blueberry Variety) | Phytochemical-poor Blueberry Variety (Olympia Blueberry Variety) | "Minimally Processed" Blueberry-rich Protein Bar | Control Beverage of Matched-nutritive Content
Number analyzed (Participants) | 18 | 18 | 18 | 18
ng/mL | 15.37 [0.43 to 63.75] | 8.44 [0.36 to 25.82] | 11.15 [0.37 to 28.17] | 6.96 [0.21 to 32.34]
Statistical Analysis 1: Comparison: Phytochemical-rich Blueberry Variety (Elliott Blueberry Variety) vs Phytochemical-poor Blueberry Variety (Olympia Blueberry Variety) vs "Minimally Processed" Blueberry-rich Protein Bar vs Control Beverage of Matched-nutritive Content; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.05, ANOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

4. Other Pre Specified Outcome: Time at Maximum Concentration [Tmax] of (Poly)Phenolic Metabolites in Serum Between the Treatments
Description: Concentration of 185 (poly)phenolic metabolites in serum was measured after consumption of the treatments using broad spectrum metabolomic analysis via UPLC-MS/MS (ultra-performance liquid chromatography coupled with tandem mass spectrometry). The time at maximum serum concentration [Tmax] of each (poly)phenolic metabolite in serum was calculated per participant and treatment using concentration and time data in the software Phoenix WinNonlin (version 8.3, Certara). Then, it was averaged across participants per treatment and per metabolite, and further averaged across metabolites. Data reported for each treatment represents the mean of the means of Tmax across (poly)phenolic metabolites.
Time Frame: as for outcome 2
Population: All participants who completed all study visits. This analysis was pre-specified to only report data for (poly)phenolic metabolites that displayed treatment-by-time, treatment, and time effects (p < 0.05) in serum concentration (i.e., 20 (poly)phenolic metabolites). Mean of the means of Tmax across metabolites is reported per treatment.
Measure: Mean (Full Range); unit: hour
Arm/Group | Phytochemical-rich Blueberry Variety (Elliott Blueberry Variety) | Phytochemical-poor Blueberry Variety (Olympia Blueberry Variety) | "Minimally Processed" Blueberry-rich Protein Bar | Control Beverage of Matched-nutritive Content
Number analyzed (Participants) | 18 | 18 | 18 | 18
hour | 6.35 [3.65 to 10.34] | 6.96 [2.91 to 12.35] | 7.70 [2.48 to 16.66] | 9.96 [1.33 to 19.83]
Statistical Analysis 1: Comparison: Phytochemical-rich Blueberry Variety (Elliott Blueberry Variety) vs Phytochemical-poor Blueberry Variety (Olympia Blueberry Variety) vs "Minimally Processed" Blueberry-rich Protein Bar vs Control Beverage of Matched-nutritive Content; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.05, ANOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From participant enrollment to study completion (3.9 ± 1.7-mo period).
Groups:
- a Phytochemical-rich Blueberry Variety (Elliott Blueberry Variety): Single-time consumption of 150 g phytochemical-rich blueberry per participant.
  a non-traditional (i.e., not typically available in the supermarket) blueberry cultivar bred using natural plant breeding techniques and established as having enhanced nutritive value: 150 g of a non-traditional (i.e., not typically available in the supermarket) blueberry cultivar bred using natural plant breeding techniques and established as having enhanced nutritive value.
  Dietary restrictions will be observed (i.e. avoidance of food or supplements containing berry phytonutrients) for 7 days before each arm visit and throughout the study days.
- a Phytochemical-poor Blueberry Variety (Olympia Blueberry Variety): Single-time consumption of 150 g phytochemical-poor blueberry per participant.
  a standard commercially available blueberry variety (i.e., cultivar): 150 g of a standard commercially available blueberry variety (i.e., cultivar).
  Dietary restrictions will be observed (i.e. avoidance of food or supplements containing berry phytonutrients) for 7 days before each arm visit and throughout the study days.
- a "Minimally Processed" Blueberry-rich Protein Bar: Single-time consumption of blueberry-rich protein bar matched for 150 g blueberry phytochemicals.
  a "minimally processed" blueberry-rich protein bar: A "minimally processed" blueberry-rich protein bar matched to the phytonutrient content of the 150 g of the non-traditional blueberry.
  Dietary restrictions will be observed (i.e. avoidance of food or supplements containing berry phytonutrients) for 7 days before each arm visit and throughout the study days.
- a Blueberry Control Beverage of Matched-nutritive Content: Single-time consumption of control beverage matched for the macronutrient content of the blueberry-rich protein bar.
  a control beverage of matched-nutritive content: The matched nutritive content of the blueberry-rich protein bar will be dissolved in whey protein
  Dietary restrictions will be observed (i.e. avoidance of food or supplements containing berry phytonutrients) for 7 days before each arm visit and throughout the study days.
Arm/Group | a Phytochemical-rich Blueberry Variety (Elliott Blueberry Variety) | a Phytochemical-poor Blueberry Variety (Olympia Blueberry Variety) | a "Minimally Processed" Blueberry-rich Protein Bar | a Blueberry Control Beverage of Matched-nutritive Content
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/18

LIMITATIONS AND CAVEATS:
Some limitations in this study include the lack of a software to evaluate background diet, and lack of measurement of composition of the protein bars. Further, compliance to a diet low in (poly)phenols (but not polyphenol-free) was evaluated through food intake logs and a strictly controlled and (poly)phenol-free diet is only feasible in a metabolic ward/domicile study design, which is relatively rare for (poly)phenol interventions. Also, we cannot account for nonreported noncompliance events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/06/NCT04175106/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-25): https://cdn.clinicaltrials.gov/large-docs/06/NCT04175106/SAP_001.pdf
  • Informed Consent Form: Informed Consent Form (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT04175106/ICF_002.pdf
  • Informed Consent Form: Informed Consent Addendum (2020-08-04): https://cdn.clinicaltrials.gov/large-docs/06/NCT04175106/ICF_003.pdf